CLINICAL TRIAL: NCT02072733
Title: Oncogeriatric Intervention and Follow-up at Home to Improve Quality of Life and the Possibility to Accomplish Cancer Treatment in Multimorbid Elderly
Brief Title: Suitability of an Organization With an Onco-geriatric Team to a Whole Region (Region Midt) of Denmark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Oncogeriatric feasibility
Record Dates: First submitted 2014-02-19; First posted 2014-02-27 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2015-12

CONDITIONS: Elderly; Cancer
Keywords: frailty; oncogeriatrics; Multidisciplinary intervention; multimorbidity; Comprehensive geriatric assessment; patients
MeSH Terms: conditions — Neoplasms; Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- geriatric assessment (Other): The intervention is individual and based on the Comprehensive Geriatric assessment (CGA) : collection of information on comorbidity, polypharmacy, physical, psychological and cognitive functions, nutrition as well as social status and support.
  The results of the CGA, the eventual medical changes and recommendations regarding e.g. initiation of nutritional supplementation, home-care referral or referral to e.g. physiotherapist will be forwarded to the general practitioner and to the oncologist in charge of the treatment
  Interventions: Other: Comprehensive geriatric assessment

INTERVENTIONS:
Other: Comprehensive geriatric assessment — Intervention is planned to be based on the findings of the geriatric assessment and could include optimizing on comorbidity, planning of physical exercise, improvement of the social situation and nutritional status.

SUMMARY:
A Feasibility study Geriatric assessment applied to patients with cancer of the head and neck, lung cancer, upper gastrointestinal cancer or colo-rectal cancer. On the day of planning the oncologic treatment Comprehensive Geriatric Assessment (CGA) will be offered to patients aged 70 years and up. Based on the CGA a tailored multidisciplinary intervention is planned with the patients. The study aims 1) to investigate if it is feasible to offer CGA to all elderly (+70 years) patients with the relevant cancer diagnoses as mentioned above in The Central Denmark Region (Region Midt) , 2) to estimate the proportion of frail, vulnerable or fit elderly cancer patients, 3) to investigate the impact of a CGA on the planned oncologic treatment intensity, and 4) to investigate the ability of CGA to predict complications to cancer treatment within a three months period.

DETAILED DESCRIPTION:
Aim:

The study aims 1)to investigate if it is feasible to offer CGA to all elderly (+70 years) patients with the relevant cancer diagnoses as mentioned above in The Central Denmark Region (Region Midt) , 2) to estimate the proportion of frail, vulnerable or fit elderly cancer patients, 3) to investigate the impact of a CGA on the planned oncologic treatment intensity and 4)to investigate the ability of CGA to predict complications to cancer treatment within a three months period.

Method:

All patients referred to the oncology Departement aged 70 years or more with cancer of the head and neck, lung cancer, upper gastrointestinal cancer or colo-rectal cancer, Living in the Central Denmark Region (Region Midt) are offered af Comprehensive Geriatric Assessment (CGA) on the day of the visit to the oncology outpatient Clinic. Prior to the first visit to the oncology department, the patients are informed that a CGA is planned..The CGA will take place at the outpatient clinic. The results of the CGA, the eventual medical changes and recommendations regarding e.g. initiation of nutritional supplementation, home-care referral or referral to e.g. physiotherapist will be forwarded to the general practitioner and to the oncologist in charge of the treatment.

Outcome:

1. The possibility of offering CGA to elderly cancer patients in a larger area, the proportion of patients offered CGA by the oncogeriatric team compared to the actual number of elderly cancer patients assessed by oncologists during a three months period.
2. The number of frail vs. vulnerable vs. fit persons is estimated from hospital records and the CGA observations. Their dependency in Activities of Daily Living (ADL) and Instrumental Activities og Daily Living (IADL), their cognitive, depressive and nutritional status and the medication problems are registered as well as the changes in patient´s medication.
3. The impact of CGA on the oncologist´s treatment plan.
4. The Complications, defined as discontinuation of treatment, hospitalization for other reasons than planned cancer treatment, or death, within the first three month following CGA.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* Patients from Central Denmark Region (Region Midtjylland)
* Lung cancer, Upper Gastrointestinal Cancer, cancer of head and neck and Colo-Rectal Cancer
* referred for assessment of treatment to the oncological department at Aarhus University Hospital.

Exclusion Criteria:

Patients referred to specialized palliative care at the first visit to the oncological outpatient clinic.

Ages: 70 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | 3 months
  Description of the proportion of patients who is available for CGA presented in percentage. Proportion of patients missed for CGA due to organisational issues or rejection to participate in the geriatric evaluation is presented in percentage.

SECONDARY OUTCOMES:
frailty status | 3 months
  Patient characteristics according to CGA status is presented in percentage

OTHER OUTCOMES:
Impact of CGA on the oncologist´s treatment plan | 3 months
  To analyse the association between the oncologist´s initial treatment plan (standard dose, reduced dose or supportive/palliative/no treatment) and the CGA conclusion (fit, vulnerable or frail) Pearson´s Chi-squared-test or Fisher´s Exact test is used.
  In a subgroup analysis on the non-agreed category data on the CGA conclusion and the oncologist´s initial treatment plan. And furthermore to compare the oncologist´s final treatment intensity to the CGA recommendations Pearson´s Chi-squared-test or Fisher´s Exact test are used
Complications | 3 months
  Description of the proportion of patients who is available for CGA presented in percentage. Proportion of patients missed for CGA due to organisational issues or rejection to participate in the geriatric evaluation is presented in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Else Marie Damsgaard, Professor, Study Chair — Geriatric Department Aarhus University Hospital Denmark
Locations (1):
- Geriatric Department Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No